CLINICAL TRIAL: NCT04505449
Title: Role of Invasive Left Heart Catheterization for Patients Suspected Heart Failure With Preserved Ejection Fraction
Brief Title: Invasive Left Heart Catheterization Registry
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeong Hoon Yang, Professor, Samsung Medical Center
Other Study IDs: LHCR
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Left Ventricular Diastolic Dysfunction
Keywords: Heart failure with preserved ejection fraction; Left ventricular end diastolic pressure; Echocardiography
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Left heart catheterization: Symptomatic patients who underwent left heart catheterization and coronary angiography.
  Interventions: Diagnostic Test: Left heart catheterization

INTERVENTIONS:
Diagnostic Test: Left heart catheterization — Patients who underwent left heart catheterization

SUMMARY:
Retrospectively enrolled suspicious of heart failure with preserved ejection fraction (HFpEF) patients who underwent left heart catheterization with the measurement of left ventricular end-diastolic pressure.

DETAILED DESCRIPTION:
Heart failure (HF) with preserved ejection fraction (HFpEF) remains a poorly understood clinical syndrome without effective targeted therapies. The clinical syndrome of HFpEF develops from a complex interaction of several risk factors such as aging, obesity, hypertension, myocardial ischemia, and arterial stiffness that cause organ dysfunction and, ultimately, clinical symptoms. Although the H2FPEF and HFA-PEFF scores have recently been proposed to estimate the probability of HFpEF in patients suffering from unexplained dyspnea, diagnosing HFpEF remains still challenging. The aim of the current registry was to evaluate the role of invasive left heart catheterization with the measurement of left ventricular end-diastolic pressure (LVEDP) in suspicious of HFpEF patients.

ELIGIBILITY:
Inclusion Criteria:

* Left ventricular ejection fraction > 50%
* Patients who had a symptom and/or signs of heart failure (dyspnea on exertion, chest discomfort, fatigue, dizziness, or ankle edema)
* Patients who underwent left heart catheterization with the measurement of left ventricular end-diastolic pressure

Exclusion Criteria:

* Left ventricular ejection fraction <50%
* Acute coronary syndrome
* More than moderate valvular heart disease
* Primary cardiomyopathies such as dilated cardiomyopathy and hypertrophic cardiomyopathy, amyloidosis
* Pulmonary arterial hypertension
* Heart transplantation
* Constrictive pericarditis
* Stress-induced cardiomyopathy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospectively enrolled symptomatic patients who underwent left heart catheterization
Sampling Method: Non-Probability Sample
Enrollment: 404 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Rates of Death or re-hospitalization due to heart failure | 10 Years

SECONDARY OUTCOMES:
Rates of All-cause death | 10 Years
Rates of Re-hospitalization due to heart failure | 10 Years
Rates of Myocardial infarction | 10 Years
Rates of Stroke | 10 Years

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Hoon Yang, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi KH, Yang JH, Seo JH, Hong D, Youn T, Joh HS, Lee SH, Kim D, Park TK, Lee JM, Song YB, Choi JO, Hahn JY, Choi SH, Gwon HC, Jeon ES. Discriminative Role of Invasive Left Heart Catheterization in Patients Suspected of Heart Failure With Preserved Ejection Fraction. J Am Heart Assoc. 2023 Mar 21;12(6):e027581. doi: 10.1161/JAHA.122.027581. Epub 2023 Mar 9. PMID 36892042